CLINICAL TRIAL: NCT05597384
Title: Assessment of Autologous Blood Marker Localization and Intraoperative Colonoscopy Localization in Laparoscopic Colorectal Cancer Surgery: a Randomized Controlled Trial
Brief Title: Assessment of Autologous Blood Marker Localization in Laparoscopic Colorectal Cancer Surgery
Acronym: ABILITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shanghaieasthospital-2022113
Record Dates: First submitted 2022-10-23; First posted 2022-10-28 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Autologous blood; Endoscopy tattooing; Preoperative localization
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Blood Marker Group (Experimental): The tattooing was performed at 24-48 hours before the surgery. When the lesion was identified by endoscopy, 2-3 ml of the patient's peripheral venous blood without heparin preparation were injected submucosally at the distal side and proximal side of the lesion using a conventional endoscopic needle without submucosal injection of normal saline.
  Interventions: Procedure: Laparoscopic colorectal cancer resection
- Intraoperative colonoscopy group (Active Comparator): Under general anesthesia with endotracheal intubation, the patient was placed in the modified lithotomy position. After routine laparoscopic exploration, CO2-insufflated intraoperative colonoscopy was performed using a flexible videocolonoscope. Upstream small bowel clamping was applied before intraoperative colonoscopy. During intraoperative colonoscopy, CO2 pneumoperitoneum was maintained by the insufflator so that the laparoscope could guide the colonoscope effectively.
  Interventions: Procedure: Laparoscopic colorectal cancer resection

INTERVENTIONS:
Procedure: Laparoscopic colorectal cancer resection — This is one of the routine procedures used for colorectal cancer resection.

SUMMARY:
Laparoscopic colorectal surgery has been proved to have similar oncological outcomes with open surgery. Due to the lack of tactile perception, surgeons may have misjudgments in laparoscopic colorectal surgery. Therefore, the accurate localization of a tumor before surgery is important, especially in the early stages of cancer. Recently, some retrospective studies reported the use of patients' autologous blood for preoperative colonic localization in colorectal cancer with successful detection by laparoscopy, but its benefits remain controversial. This study aimed to assess the accuracy and safety of autogenous blood marker localization in laparoscopic radical resection for colorectal cancer.

DETAILED DESCRIPTION:
Laparoscopic surgery has become the standard for management of colorectal cancer(CRC) with the advantages of less traumatic procedure, but similar oncological outcomes to open surgery. Due to the lack of tactile perception (haptic feedback), surgeons may have misjudgments in patients with small or flat early colon cancer, malignant polyps resected by endoscopic mucosal resection or endoscopic submucosal dissection. Therefore, the accurate localization of a tumor before surgery is important, especially in the early stages of cancer, to clarify the extent of surgical resection.

Several methods are currently being proposed and used to identify the location of tumors. These include endoscopic tattooing with India ink, indocyanine green (ICG), preoperative endoscopic metal clipping with detection using an x-ray or palpation during surgery, and intraoperative endoscopy.

Recently, some retrospective studies reported the use of patients' autologous blood for preoperative colonic localization in CRC with successful detection by laparoscopy. Autologous blood was thought a feasible and safe tattooing agent for preoperative endoscopic localization. Nonetheless, all currently available evidence comes from observational studies that are susceptible to bias. We therefore proposed to conduct this randomized controlled clinical trial to evaluate the accuracy and safety of autogenous blood marker localization in laparoscopic radical resection for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years
2. Large lateral spreading tumors that could not be treated endoscopically, serosa-negative malignant colorectal tumors (≤ cT3), and malignant polyps treated endoscopically that required additional colorectal resection.
3. The tumor is located in the colon, middle and high rectum (the lower margin of the tumor does not exceed peritoneal reflexes)
4. No distant metastasis.
5. American Society of Anesthesiology score (ASA) class I-III
6. Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
7. Written informed consent

Exclusion Criteria:

1. BMI > 35kg/m2
2. Previous history of gastrointestinal surgery that altered the gastrointestinal anatomy.
3. Pregnant or lactating women
4. Severe mental disorder
5. History of previous abdominal surgery (except cholecystectomy and appendectomy) Rejection of laparoscopic resection
6. History of cerebrovascular accident within the past six months
7. History of unstable angina or myocardial infarction within the past six months
8. History of previous neoadjuvant chemotherapy or radiotherapy
9. Comorbidity of emergent conditions like obstruction, bleeding or perforation.
10. Needing simultaneous surgery for other diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Autogenous blood marker localization was not inferior to intraoperative colonoscopy localization | From the beginning of endoscopic tattooing to the end of the surgery.
  While checking the intraperitoneal cavity at the start of the surgery, the visibility of tattooing will be first checked. After the complete resection of the colon segment, resected colon specimen will be checked the localization with autologous blood tattooing. The localization accuracy of autologous blood marker will be similar to that of intraoperative colonoscopy localization.

SECONDARY OUTCOMES:
Adverse events related to endoscopic tattooing | From the beginning of colonoscopic tattooing to 2 weeks after surgery.
  The secondary endpoint is the localization safety. Adverse events related to endoscopic tattooing, such as perforation, abscess formation, peritonitis, post-tattoo fever, post-tattoo abdominal pain, and intraperitoneal spillage of tattooing agent, were evaluated in autologous blood group.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang KH, Li JZ, Zhang HB, Hu RH, Cui XM, Du T, Zheng L, Zhang S, Song C, Xu MD, Jiang XH. Assessment of Autologous Blood marker localIzation and intraoperative coLonoscopy localIzation in laparoscopic colorecTal cancer surgery (ABILITY): a randomized controlled trial. BMC Cancer. 2023 Mar 3;23(1):204. doi: 10.1186/s12885-023-10669-w. PMID 36869328